CLINICAL TRIAL: NCT02630498
Title: The Role of Single Shot Brachial Plexus Block in Preventing Chronic Post Surgical Pain After Upper Limb Trauma Surgery
Brief Title: Preventing Chronic Post Surgical Pain After Limb Surgery
Acronym: PCPSPAULS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It was not practical to continue recruiting due to lack of human resources
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shalini Dhir, AssociateProfessor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSREB 105321
Record Dates: First submitted 2015-08-11; First posted 2015-12-15 (Estimated); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Chronic Pain
Keywords: pain; surgical; brachial plexus
MeSH Terms: conditions — Chronic Pain; Pain | interventions — Brachial Plexus Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- study (first group) (Experimental): The first group will include those who receive a single shot brachial plexus block with or without general anesthesia.
  Interventions: Procedure: Brachial plexus block
- Controlled (second group) (No Intervention): The second group will be the control group and include those patients who receive general anesthesia only, without any block whether due to the preference of patient or the surgeon.

INTERVENTIONS:
Procedure: Brachial plexus block — Patients receiving brachial plexus block for hand/arm surgery
  Arms: study (first group)

SUMMARY:
This is a non-randomized prospective study. Patients undergoing upper extremity and shoulder surgical procedures after trauma at SJHC and LHSC will be divided in to two groups. The first group will include those who receive a single shot brachial plexus (interscalene, supraclavicular, infraclavicular and axillary) block with or without general anesthesia. The second group will be the control group and include those patients who receive general anesthesia only, without any block whether due to the preference of patient or the surgeon

DETAILED DESCRIPTION:
This is a non-randomized prospective study. Patients undergoing upper extremity and shoulder surgical procedures after trauma at SJHC and LHSC will be divided in to two groups. The first group will include those who receive a single shot brachial plexus (interscalene, supraclavicular, infraclavicular and axillary) block with or without general anesthesia. The second group will be the control group and include those patients who receive general anesthesia only, without any block whether due to the preference of patient or the surgeon. Patients will not be randomized for this study because regional anesthesia is proven to reduce acute postoperative pain and reduce the need for opioids. However, investigators will involve all patients who meet the inclusion criteria and give consent to participate in this study within the period of study between September 1st 2015 and February 28th 2017 (18 months). The block is usually performed with ultrasound guidance by the block Room team at both sites (consultant, fellow and resident). Block success will be checked and documented. Ropivacaine is the standard local anesthetic used in the block room at LHSC (University Hospital) and SJHC. However, the type of local anesthetics and the total volume are difficult to be standardized for all patients in this study, so it will be neglected during analysis. The block room at SJHC and LHSC perform around 100 blocks per month. Thirty percent of these blocks are for upper limb procedures. The same number of patients undergoes these procedures with no blocks at both SJHC and LHSC. Investigators expect to involve around 100 patients in each arm during the study period. All patients will be followed up for 6 months through filling a questionnaire and Brief Pain Inventory (BPI), which assess pain score and pain interference scale. The follow up will be through mail and /or phone call. Sample Size There is no previous study data provided the prevalence of CPSP in similar surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Trauma patient undergoing orthopedic surgery for upper extremity or shoulder
2. Age >18 and < 75 years
3. Both males and females
4. Understand English (reading, writing and speaking)
5. Patient gives a written consent for being involved in this study

Exclusion Criteria:

1. Patient with any sort of chronic pain including fibromyalgia
2. Patient using opioids for >90 days
3. Patient who had an associated injury related to the trauma apart from that limb
4. Patient who need more than one surgery to fix the problem
5. Patient diagnosed with major depression
6. Failed or partially effective block
7. Bilateral surgical intervention

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Chronic Post Surgical Pain | Upto six months

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Dhir, FRCPC, Principal Investigator — LHSC
Locations (2):
- Canada (2):
  - St. Joseph's Hospital, London, Ontario
  - LHSC, SJHC, Western University, London, Ontario

IPD SHARING:
Plan to Share IPD: No